CLINICAL TRIAL: NCT06276556
Title: A Multicenter, Double-blind, Phase 2b/3 Extension Study to Assess the Safety and Efficacy of ABP-671 in Participants With Gout Who Completed the Double-blind Treatment Period in Study ABP-671-301
Brief Title: Extension Study of ABP-671 in Participants With Gout
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: For business consideration, a new long-term safety study will be conducted in the next new pivotal studies.
Sponsor: Atom Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABP-671-302
Record Dates: First submitted 2024-02-12; First posted 2024-02-26 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2024-08

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ABP-671 (Experimental)
  Interventions: Drug: ABP-671
- Allopurinol (Active Comparator)
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: ABP-671 — Participants who were randomized to any of the ABP-671 treatment groups in Part 1 or Part 2 of Study ABP-671-301 will continue to receive the same dose level and dosing regimen during the Treatment Period of this Extension Study.
  Participants who were randomized to receive placebo in Part 1 or Part 2 of Study ABP-671-301 will receive ABP-671 during the Treatment Period of the Extension Study.
  Arms: ABP-671
Drug: Allopurinol — Participants who were randomized to receive allopurinol in Part 1 of Study ABP-671-301 will continue to receive allopurinol during the Treatment Period of the Extension Study.
  Arms: Allopurinol

SUMMARY:
The primary objectives of this study are to assess the safety, tolerability, and efficacy of ABP-671 in lowering serum uric acid (sUA) in participants with gout who roll over from Study ABP-671-301 after they complete the double-blind 28-week Treatment Period of Part 1 (Phase 2b) or Part 2 (Phase 3).

ELIGIBILITY:
Inclusion Criteria:

* Must have completed the double-blind Treatment Period in Study ABP-671-301 (Part 1 or Part 2) and are actively receiving and tolerating the study drug up to the Week 28 visit in Study ABP-671-301

Exclusion Criteria:

* Has a new medical or psychological condition that, in the opinion of the Investigator and/or Medical Monitor, might create undue risk to the participant, interfere with the participant's ability to comply with the protocol requirements to complete the Extension Study, or potentially compromise the results or interpretation of the Extension Study.
* Is planning to become pregnant or breastfeed during the study or within ≤30 days after the last dose of the study drug.
* Is intolerant or unwilling to take colchicine or naproxen.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who achieve serum uric acid (sUA) levels <6.0 mg/dL (<0.360 mmol/L) | Week 26
Incidence of treatment-emergent adverse events (Safety and Tolerability) | Week 26
  Incidence of treatment-emergent adverse events (TEAEs), including AEs of special interest (AESIs), serious AEs (SAEs), and AEs leading to study treatment discontinuation

SECONDARY OUTCOMES:
Proportion of participants who achieve sUA levels <5.0 mg/dL (<0.300 mmol/L) | Week 26

CONTACTS AND LOCATIONS:
Locations (54):
- United States (33):
  - Alliance for Multispecialty Research, Tempe, Arizona
  - Tucson Neuroscience Research, LLC, Tucson, Arizona
  - Anaheim Clinical Trials (Cenexel ACT), Anaheim, California
  - Center for Clinical Trials of Sacramento, Sacramento, California
  - Access Research Institute, Brooksville, Florida
  - Nature Coast Clinical Reasearch, Crystal River, Florida
  - JY Research Institute Inc., Cutler Bay, Florida
  - Accel Clinical Research Site, DeLand, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - A & D Doctor Center, Miami, Florida
  - Bioclinical Research Alliance, Miami, Florida
  - Cordova Research Institute, Miami, Florida
  - Century Research LLC, Miami, Florida
  - ITB Research, Miami, Florida
  - Combined Research Orlando Phase I-IV, Orlando, Florida
  - New Horizons Research, Palmetto Bay, Florida
  - Advanced Clinical Research of Atlanta, Atlanta, Georgia
  - Centricity Research, Columbus, Georgia
  - Alliance for Multispecialty Research, LLC., Newton, Kansas
  - DelRicht Research, New Orleans, Louisiana
  - AMR, New Orleans, Louisiana
  - Annapolis Internal Medicine/CCT Research, Annapolis, Maryland
  - DelRicht Research of Gulfport, Gulfport, Mississippi
  - Quality Clinical Research, Inc, Omaha, Nebraska
  - Santa Rosa Medical Center, Las Vegas, Nevada
  - Inspire Santa Fe Medical Group, Santa Fe, New Mexico
  - OnSite Clinical Solutions, Salisbury, North Carolina
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - ClinSearch, Chattanooga, Tennessee
  - Medical Care/CCT, Elizabethton, Tennessee
  - PanAmerican Clinical Research, LLC, Brownsville, Texas
  - Quality Research Inc., San Antonio, Texas
  - Worldwide Clinical Trials, San Antonio, Texas
- Australia (6):
  - Paratus Clinical Research Western Sydney, Blacktown, New South Wales
  - Emeritus Research Sydney, Botany, New South Wales
  - Paratus Clinical Research Central Coast, Kanwal, New South Wales
  - A R Houston Medical Pty Ltd, Kippa-Ring, Queensland
  - Emeritus Research Melbourne, Camberwell, Victoria
  - Austin Health - Repatriation Hospital, Heidelberg, Victoria
- Georgia (6):
  - New Hospitals, Tbilisi
  - Evex Hospitals Caraps Medline, Tbilisi
  - Aversi Clini, Tbilisi
  - The First Medical Center, Tbilisi
  - Academician Vakhtang Bochorishvili Clinic, Tbilisi
  - Innova, Tbilisi
- Guatemala (4):
  - Clinical Research Center (CRC), Guatemala City
  - Clínica Médica Especializada en Medicina Interna y Reumatología (CREER), Guatemala City
  - Clínica Médica Especializada en Medicina Interna y Reumatología, Guatemala City
  - Clínica Médica Especializada en Medicina Interna, Guatemala City
- Taiwan (5):
  - Buddhist Dalin Tzu Chi General Hospital, Chiayi City
  - Chang Gung Memorial Hospital CGMH, Kaohsiung City
  - Chung Shan Medical Univ. Hospital, Taichung
  - Cheng-Shin General Hospital, Taipei
  - Chang Gung Memorial Hospital LinKou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No